CLINICAL TRIAL: NCT00414713
Title: Randomized and Controlled Clinical Trial of Transfusional Requirements in Patients With Acute Gastrointestinal Bleeding.
Brief Title: Transfusion Requirements in Gastrointestinal (GI) Bleeding
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/02/102/1729 HCSCSP
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-12

CONDITIONS: Upper Gastrointestinal Bleeding; Cirrhosis; Portal Hypertension
Keywords: Upper GI bleeding; Cirrhosis; Portal hypertension; Non-variceal bleeding; Transfusion
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Fibrosis; Hypertension, Portal | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Regular transfusion
  Interventions: Procedure: red blood cell transfusion
- 2 (Active Comparator): Restricted transfusion
  Interventions: Procedure: red blood cell transfusion

INTERVENTIONS:
Procedure: red blood cell transfusion — red blood cell transfusion

SUMMARY:
Recently it has been suggested that a restrictive transfusion of units of Red Cells (URC) may improve the outcome of ICU patients with anemia. Furthermore, it has been suggested that the transfusion of URC may be deleterious for the hemostatic process of bleeding lesions, which suggest that a restrictive transfusion may be valuable in patients which gastrointestinal bleeding. Transfusion of URC may also increase portal pressure which may be detrimental to control acute portal hypertensive bleeding.

The aim of the present study is to assess whether a restrictive transfusions may improve the outcome of patients with acute nonvariceal gastrointestinal bleeding, and also whether such a restrictive strategy may improve the outcome of bleeding episodes related with portal hypertension.

The study will be carried out with a prospective, randomized and controlled design comparing the restrictive transfusion strategy with the usual nonrestrictive transfusional strategy. Overall 860 patients will be included; 430 in each group.

The main outcome measure will be survival. All deaths occurred within the 30 days after admission, will be considered. Secondary outcomes will include rebleeding and complications related to treatment, and related to the bleeding episode itself. Portal pressure will be measured to assess the influence of the transfusions strategy on fluctuations of this parameter, and the relationship with the clinical course of bleeding episode.

The study will be performed at the Bleeding Unit of our hospital during a period of 3 years.

DETAILED DESCRIPTION:
HYPOTHESIS

At the present time there does not exist established criteria to decide when it is necessary a blood transfusion in a patient with digestive hemorrhage, neither which should be the red cells concentrates (RBC) amount that the most of the patients will need.

In clinical studies made in critical patients undergoing a by-pass coronary surgery, the strategy of restrictive transfusion showed results similar to the one obtained with more liberal strategies, even with an improvement of the survival and a smaller rate of complications related to transfusion.

In animal models of GI bleeding (and also in human studies in the traumatic hemorrhage), precocious or vigorous transfusion made hemostasia more difficult. Also an increase in the rate of rebleeding has been observed, suggesting that arterial hypotension combined with hypovolemia aid hemostasia, stabilize the clot. It leads to diminish by itself the rebleeding rate.

In the same way, in patients with portal hypertension associated hemorrhage, aggressive replacement of volemia causes increases on the portal pressure, and that could lead in a condition of bigger difficulty for the control of the hemorrhage and greater rate of recidiva.

On the other hand, potential complications associated with the transfusion would be seen potentially reduced.

Our randomized prospective study tries to demonstrate that the use of a restrictive strategy in the sanguineous transfusion in patients with acute GI upper bleeding can be at least as beneficial than the habitually used.

Moreover, restricted transfusion in these patients could improve short term survival, as well as a smaller rate transfusion-related or rebleeding.

In portal hypertension related hemorrhage, restricted transfusion could avoid fluctuations of portal pressure caused by transfusion during the acute phase of hemorrhage, which could favor hemostasia in these patients.

OBJECTIVES

The main objective is to evaluate if restrictive transfusion criterion in patients with acute upper GI hemorrhage can maintain the rates of survival obtained using habitual transfusion criteria, or to even improve them.

The more important secondary targets consist in evaluating if these restrictive transfusional parameters are also accompanied by a better control of the hemorrhage, and also to evaluate if this is accompanied by a smaller rate of complications.

Other additional objectives would be:

* Effect on changes in portal pressure and its correlation with the clinical evolution.
* Hospital stay and estimation of economic cost.

STUDY DESIGN

Ours is a prospective, randomized and controlled study, in which patients with acute upper GI bleeding will be randomized into two groups of transfusional RBC treatment with:

Group 1 (of restricted transfusion), that constitutes the training group: they will receive UCH transfusion when the hemoglobin descends below 70 G/L, to maintain values of hemoglobin of 70 to 90 G/L.

Group 2 (of habitual transfusion), that constitutes the group control: they will receive transfusion according to habitual practice, when the hemoglobin descends below 90 G/L, to maintain values of hemoglobin of 90 to 110 G/L.

Randomization will be made by means of a closed opaque envelope that will contain the treatment option that will have been obtained by means of a listing of random numbers generated by computer.

The patients will be randomized as soon as the inclusion criteria/exclusion has been verified.

Randomization will be stratified according to the origin of the hemorrhage (related to portal hypertension or not).

NUMBER OF PREDICTED SUBJECTS AND JUSTIFICATION:

430 patients in every group will be required (860 altogether), to objective a mortality reduction of 5%, with a global expected mortality secondary to GI bleeding at the control group of 10%, with a type I error of 5% and a type II error of 20%.

280 patients in each group will be required (560 altogether) to objective a difference of 6%, with the detailed parameters.

An expected period of 3 years to include this

ELIGIBILITY:
Inclusion Criteria:

* All patients with acute upper GI hemorrhage who do not have any criterion of exclusion.

Exclusion Criteria:

* < 18 years old.
* Pregnancy.
* Negative of the patient to receive transfusions.
* Negative of the patient to participate in the study.
* Patients with therapeutic restrictions (as terminally ill patients).
* Previous recent surgery requiring transfusion.
* Recent (less than 90 days) or unstable acute myocardic ischemia. Peripheral vasculopathy with secondary.
* To have been included in this same study in the 30 previous days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Estimated)
Dates: Start 2002-10; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Mortality at the 45th day | 45 days

SECONDARY OUTCOMES:
Mortality at the 7th and 45th day | 45 days
Rebleeding | 45 days
Transfusion requirements | 45 days
Liquids requirements | 45 days
Portal pressure changes | 7 days
Complications | 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Càndid Villanueva, DR, Principal Investigator — HSCSP
Locations (1):
- Unidad de Sangrantes, HSCSP, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Villanueva C, Colomo A, Bosch A, Concepcion M, Hernandez-Gea V, Aracil C, Graupera I, Poca M, Alvarez-Urturi C, Gordillo J, Guarner-Argente C, Santalo M, Muniz E, Guarner C. Transfusion strategies for acute upper gastrointestinal bleeding. N Engl J Med. 2013 Jan 3;368(1):11-21. doi: 10.1056/NEJMoa1211801. PMID 23281973